CLINICAL TRIAL: NCT03912363
Title: Intrapartum Glycemic Control With Insulin Infusion Versus Rotating Fluids: Randomized Controlled Trial (RCT)
Brief Title: Intrapartum Glycemic Control With Insulin Infusion Versus Rotating Fluids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0502
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Type II Diabetes Mellitus; Gestational Diabetes Mellitus
Keywords: intrapartum; glycemic control; diabetes; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rotating fluids (Active Comparator): Rotating fluids protocol will be initiated at the time of admission to Labor and Delivery.
  Interventions: Other: Rotating fluids protocol
- Insulin infusion (Active Comparator): Insulin infusion protocol will be initiated at the time of admission to Labor and Delivery.
  Interventions: Other: Insulin infusion protocol

INTERVENTIONS:
Other: Rotating fluids protocol — IV fluids at a rate of 100-150 ml/hr will be administered:
  * For blood glucose < 100 mg/dL or less: IV fluids with 5% dextrose
  * For blood glucose between 101-140 mg/dL: IV fluids without 5% dextrose
  * For blood glucose > 140 mg/dL on two consecutive occasions: insulin infusion protocol (Study arm 2)
  Arms: Rotating fluids
Other: Insulin infusion protocol — Regular insulin at 1 unit/ml AND IV fluids at a rate of 100-150 ml/hr will be administered:
  * For blood glucose < 80 mg/dL: No insulin AND IV fluids with 5% dextrose
  * For blood glucose 80-100 mg/dL: Insulin at 0.5 U/hr AND IV fluids with 5% dextrose
  * For blood glucose 101-140 mg/dL: Insulin at 1.0 U/hr AND IV fluids with 5% dextrose
  * For blood glucose 141-180 mg/dL: Insulin at 1.5 U/hr AND IV fluids with 5% dextrose
  * For blood glucose 181-220 mg/dL: Insulin at 2.0 U/hr AND IV fluid without dextrose
  * For blood glucose > 220 mg/dL: Insulin at 2.5 U/hr AND IV fluids without dextrose
  Arms: Insulin infusion

SUMMARY:
This study will determine whether rotating intravenous (IV) fluid is better than receiving insulin to control a baby's blood sugar after delivery in laboring women with diabetes. A computer will choose the method of controlling the participant's blood sugar while they are in labor.

DETAILED DESCRIPTION:
Diabetes complicates 6-9% of all pregnancies. Of those pregnancies, 90% of pregnant diabetics have gestational diabetes mellitus (GDM), while the remainder of patients have pre-existing diabetes mellitus (DM). Maternal hyperglycemia has a negative impact on maternal and fetal/neonatal health. Adverse neonatal outcomes include birth injuries, respiratory distress, and metabolic derangements such as hypoglycemia. The incidence of neonatal hypoglycemia is higher in pregnancies complicated by pre-existing DM (24-48%) when compared to patients with GDM (16-19%).

Neonatal hypoglycemia causes immediate and long-term morbidity. Treatment of hypoglycemia may require admission to the Neonatal Intensive Care Unit (NICU). The severity and duration of neonatal hypoglycemia raises concern for permanent neurologic damage to the neonate. Even transient episodes of neonatal hypoglycemia have been associated with neurodevelopmental impairment. It is imperative that measures be taken in diabetic mothers (both pre-existing and gestational) to minimize the risk of neonatal hypoglycemia. While antepartum maternal glucose control remains an important factor in preventing neonatal complications, prevention of maternal hyperglycemia during the intrapartum period has been shown to reduce the risk of neonatal hypoglycemia.

Therapies utilized for maternal intrapartum glycemic control across academic centers in the United States include the use of insulin and rotation of intravenous (IV) fluids. Although used in clinical practice for intrapartum glycemic control, the impact of rotating IV fluids on neonatal blood glucose is unknown. The potential for using rotating IV fluids to control intrapartum blood glucose has several advantages over using insulin for optimization of blood glucose. There is minimal risk of maternal hypoglycemia using IV fluids when compared to insulin therapy. There is also less risk of medication error. IV fluids are easily administered as they do not require separate peripheral access and are easily accessible on a Labor and Delivery (L&D) unit.

The investigators propose a randomized controlled trial (RCT) to assess the effect of maternal intrapartum glycemic control with rotating IV fluids compared to insulin infusion on neonatal blood glucose levels within two hours of birth. The investigators hypothesize neonates born to mothers managed by rotating fluids will have higher neonatal blood glucose levels (closer to normal range) within two hours of birth compared to neonates born to mothers managed by insulin infusion.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with Type II diabetes mellitus or GDM controlled with insulin and/or hypoglycemic medication (GDMA2)
* Singleton pregnancies
* Gestational age between 37 0/7 weeks and 40 0/7 weeks
* Planned delivery at a Geisinger Medical Center (GMC) or Geisinger Wyoming Valley (GWV)
* English or Spanish speaking
* Anticipated delivery at ≥ 4 hours from randomization (e.g., cervical dilation at ≤ 7 cm at time of randomization)

Exclusion Criteria:

* Women with Type 1 diabetes mellitus or use of insulin pump
* Evidence of diabetic ketoacidosis at time of admission for delivery
* Multifetal gestation
* Gestational age < 37 0/7 weeks or > 40 0/7 weeks
* Non-English or Non-Spanish speaking
* Anticipated delivery < 4 hours from randomization (e.g., cervical dilation > 7 cm at time of randomization, first cesarean delivery of the day)
* Oral corticosteroid use within 48 hours of planned delivery
* Antenatal corticosteroid use within 7 days of admission for delivery
* Delivery planned outside of GMC or GWV
* Fetal demise
* Prenatal diagnosis of lethal fetal anomaly
* Active infection or immunocompromised state (e.g., HIV/AIDS, active malignancy, use of immunosuppressant medication) at time of admission for delivery

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Neonatal blood glucose value | Within 2 hours of life
  Neonatal blood glucose value from birth to 2 hours of life

SECONDARY OUTCOMES:
Mean neonatal blood glucose value | First 24 hours of life
  Average of neonatal blood glucose values from birth to 24 hours of life
Incidence of maternal hypoglycemia | During labor (average time 24 hours)
  Blood glucose value < 50 mg/dL without symptoms OR Blood glucose value < 70 mg/dL with symptoms such as perspiration, palpitations, tremor, weakness, anxiety
Mean intrapartum maternal blood glucose value | During labor (average time 24 hours)
  Average of maternal blood glucose values during labor
Maternal blood glucose value before delivery | Within one hour of delivery
  Blood glucose value
Incidence of composite neonatal outcome | First 24 hours of life until discharge (average time 21 days)
  Neonatal hypoglycemia, NICU admission, neonatal hyperbilirubinemia, and neonatal respiratory distress syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Paglia, MD, PhD, Principal Investigator — Geisinger Clinic
Locations (2):
- United States (2):
  - Geisinger, Danville, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania

REFERENCES:
- [Background] DeSisto CL, Kim SY, Sharma AJ. Prevalence estimates of gestational diabetes mellitus in the United States, Pregnancy Risk Assessment Monitoring System (PRAMS), 2007-2010. Prev Chronic Dis. 2014 Jun 19;11:E104. doi: 10.5888/pcd11.130415. PMID 24945238
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 201: Pregestational Diabetes Mellitus. Obstet Gynecol. 2018 Dec;132(6):e228-e248. doi: 10.1097/AOG.0000000000002960. PMID 30461693
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Rosenberg VA, Eglinton GS, Rauch ER, Skupski DW. Intrapartum maternal glycemic control in women with insulin requiring diabetes: a randomized clinical trial of rotating fluids versus insulin drip. Am J Obstet Gynecol. 2006 Oct;195(4):1095-9. doi: 10.1016/j.ajog.2006.05.051. Epub 2006 Aug 8. PMID 16893507
- [Background] Golde SH, Good-Anderson B, Montoro M, Artal R. Insulin requirements during labor: a reappraisal. Am J Obstet Gynecol. 1982 Nov 1;144(5):556-9. doi: 10.1016/0002-9378(82)90227-7. PMID 6753588